CLINICAL TRIAL: NCT01163721
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group Exploratory Study to Access the Metabolic Effects of Ranolazine When Added to Ongoing Non-Insulin Antidiabetic Therapy in Subjects With Type 2 Diabetes Mellitus
Brief Title: Exploratory Study to Access the Metabolic Effects of Ranolazine in Subjects With Type 2 Diabetes Mellitus When Added to Ongoing Non-insulin Antidiabetic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-259-0107
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; T2DM; Ranolazine; Ranexa; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Experimental): Participants were randomized to receive ranolazine for 12 weeks.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Participants were randomized to receive placebo to match ranolazine for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine ER 1000 mg (two 500 mg tablets) administered orally twice daily
  Other Names: Ranexa®
  Arms: Ranolazine
Drug: Placebo — Placebo to match ranolazine administered orally twice daily
  Arms: Placebo

SUMMARY:
This study enrolled participants with inadequately controlled type 2 diabetes mellitus (T2DM) despite non-insulin antidiabetic therapy in addition to diet and exercise, and would have benefited from additional control of blood glucose levels. The study assessed the metabolic effects of ranolazine, including its effect in lowering glycosylated hemoglobin A1c (HbA1c), and lowering glucose while fasting, and following a meal (postprandial).

Participants were randomized in a 1:1 ratio to receive ranolazine or placebo, and were stratified by HbA1c ≤ 7.5% or > 7.5%. Enrollment was to include no more than two-thirds of participants with baseline HbA1c ≤ 7.5%. Other than glucose values, efficacy endpoint results remained blinded during the study; for safety purposes, the investigator was to be alerted of severe hyperglycemia or hypoglycemia.

Participants were instructed to maintain logs of their physical activity/exercise (Subject Activity Assessment) and study drug dosing (Dosing Log).

ELIGIBILITY:
Inclusion Criteria:

* Participant with T2DM on stable non-insulin antidiabetic therapy in addition to diet and exercise
* Body mass index (BMI) ≥ 25 kg/m^2 and ≤ 40 kg/m^2
* HbA1c 7 - 11%
* Ability and willingness to maintain a complete and accurate Subject Activity Log during the course of the trial
* Female of child-bearing potential must have agreed to use effective methods of contraception
* Ability to understand and willing to sign written informed consent

Exclusion Criteria:

* Type 1 Diabetes Mellitus (T1DM)
* T2DM with history of or current insulin therapy. Prior use during pregnancy or gestational diabetes was acceptable.
* History of ketoacidosis or ketosis-prone diabetes
* Clinically significant complications of diabetes that in the judgment of the investigator would have made participant unsuitable to participate in this trial
* History of a severe episode of hypoglycemia
* Change in non-insulin antidiabetic therapy in addition to diet and exercise < 2 months prior to screening
* Any clinically significant cardiovascular event < 2 months prior to screening
* Clinically significant, inadequately controlled or unstable hypertension
* Hospitalization < 2 months prior to screening
* Major surgery < 3 months prior to screening
* Weight loss medication (prescription or non-prescription) < 2 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - AMCR Institute, Escondido, California
  - National Research Institute (NRI), Los Angeles, California
  - SeaView Research Inc., Miami, Florida
  - Orlando Clinical Research Center (OCRC), Orlando, Florida
  - Midwest Institute For Clinical Research Inc. (MICR), Indianapolis, Indiana
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Rochester Clinical Research (RCR), Rochester, New York
  - Cetero Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with type 2 diabetes mellitus (T2DM) were enrolled in a total of 9 study sites in the United States. The first participant was screened on 22 June 2010. The last participant observation was on 15 November 2010.
Pre-assignment Details: The Safety Analysis Set (n = 80) includes participants who were randomized in the study and received at least one dose of study drug. The Full Analysis Set (n = 79) includes participants who were randomized in the study and received at least one dose of study drug, and had at least one post-baseline efficacy measurement.
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 39 | 41
Completed | 31 | 29
Not Completed | 8 | 12
Not completed — Adverse Event | 5 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 39 | 41 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (10.1) | 58 (9.1) | 58 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 23 | 25 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 28 | 53
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33 | 39 | 72
  Black | 5 | 1 | 6
  Other | 1 | 1 | 2
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c in blood] | 8.41 (1.078) | 8.51 (1.163) | 8.46 (1.117)
2-hour Postprandial Glucose [Mean (Standard Deviation); unit: mg/dL] — 2-hour postprandial serum glucose was defined as the average of serum glucose measurement at 120 minutes and 125 minutes following a meal.
  mg/dL | 253.1 (57.37) | 271.5 (87.67) | 262.5 (74.57)
Fasting Serum Glucose [Mean (Standard Deviation); unit: mg/dL] — Fasting serum glucose was measured following an overnight fast.
  mg/dL | 153.7 (43.05) | 172.7 (52.20) | 163.4 (48.60)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: HbA1c is a blood test to measure blood sugar control over the prior 3-month period. The last observation carried forward (LOCF) method was used: the last observed post-baseline measurements prior to Week 12 carried forward for participants with no available Week 12 values. Participants were summarized according to the actual treatment received regardless of the allocated treatment.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c in blood
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 39 | 39
percent of HbA1c in blood | -0.61 (0.142) | -0.08 (0.142)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Assuming a common standard deviation of 1.1%, 60 evaluable participants would provide 93% power to detect a statistically significant -1.0% difference in change from baseline HbA1c at Week 12 between ranolazine and placebo (2-sided alpha = 0.05). 80 participants were randomized to ensure at least 60 evaluable participants; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is from an Analysis of Covariance (ANCOVA) model with treatment as factor and baseline HbA1c value as covariate. Due to the exploratory nature of this study, there were no adjustments for multiplicity; difference in least squares mean (LSM) = -0.53, 95% CI 2-sided [-0.93 to -0.13], Standard Error of Mean 0.200

2. Primary Outcome: Change From Baseline in 2-hour Postprandial Serum Glucose at Week 12 Following a Standardized Meal
Description: 2-hour postprandial serum glucose was defined as the average of serum glucose measurement at 120 minutes and 125 minutes following a standardized meal. The LOCF method was used. Participants were summarized according to the actual treatment received regardless of the allocated treatment.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 35 | 36
mg/dL | -26.6 (9.88) | -11.2 (9.63)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.234, ANCOVA — P-value is from an ANCOVA model with treatment and baseline HbA1c stratification as factors and baseline value as covariate; difference in LSM = -15.4, 95% CI 2-sided [-41.0 to 10.2], Standard Error of Mean 12.83

3. Primary Outcome: Change From Baseline in Fasting Serum Glucose at Week 12
Description: Serum glucose was measured following an overnight fast. The LOCF method was used. Participants were summarized according to the actual treatment received regardless of the allocated treatment.
Time Frame: Baseline to Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 39 | 40
mg/dL | 2.0 (7.21) | 4.5 (6.83)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority or Other; p = 0.794, ANCOVA — [p-value comment as in outcome 2, analysis 1]; difference in least squares mean (LSM) = -2.5, 95% CI 2-sided [-21.1 to 16.2], Standard Error of Mean 9.38

ADVERSE EVENTS:
Time Frame: Baseline through Week 12
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/41
Other Adverse Events (participants affected / at risk) | 12/39 | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=39) | Placebo (N=41)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=39) | Placebo (N=41)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Headache (Nervous system disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Asthenia (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years